CLINICAL TRIAL: NCT00505934
Title: Open-label, Single-arm, Multi-center, Pharmacokinetic, Safety and Tolerability Study of Levetiracetam Intravenous Infusion in Children (1 Month- 4 Years Old) With Epilepsy
Brief Title: Open-label Study of Levetiracetam Intravenous Infusion in Children (1 Month-4 Years Old) With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01275; 2007-003517-13 (EudraCT Number)
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Child; Levetiracetam; Keppra®; Infusion; Intravenous
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Intravenous 100 mg/mL, twice a day, maximum of 4 days
  Subjects on oral levetiracetam at study entry receive the same intravenous (IV) dosage (mg-for-mg) to their oral dose within the following dose range, calculated on the basis of their age and weight:.
  * Ages ≥ 1 month to < 6 months: 14 mg/kg/day (7 mg/kg twice daily) to 42 mg/kg/day (21 mg/kg/day twice daily);
  * Ages ≥ 6 months to < 4 years: 20 mg/kg/day (10 mg/kg twice daily) to 60 mg/kg/day (30 mg/kg/day twice daily).
  For subjects not taking levetiracetam oral solution prior to entering the study, the intravenous (IV) dosage corresponded to their age and weight as follows:
  * Ages ≥ 1 month to < 6 months: 14 mg/kg/day (7 mg/kg twice daily).
  * Ages ≥ 6 months to < 4 years: 20 mg/kg/day (10 mg/kg twice daily).
  Other Names: Keppra®; ucb L059

SUMMARY:
Keppra injection is approved in the US as adjunctive therapy in the treatment of partial onset seizures in adults with epilepsy. The objective of the current study is to assess the safety, tolerability, and pharmacokinetics, of this formulation in children aged 1 month to 4 years.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the safety and tolerability of levetiracetam intravenous 15-minute infusion administered every 12 hours, either as adjunctive treatment or monotherapy in children (1 month to 4 years old) with epilepsy (except status epilepticus), either after switching from the equivalent levetiracetam oral dose administration or as a new antiepileptic treatment.

The evaluation period was to be considered as one complete set of 4 pharmacokinetic (PK) samples for a maximum of 4 days;

For children already taking levetiracetam oral solution prior to entering the study, the levetiracetam intravenous (LEV IV) dose will be equivalent (mg-for-mg) to their oral dose (always in twice daily regimen) within the following dose range, calculated on the basis of their age and weight:

* Children ≥ 1 month to < 6 months: 14 mg/kg/day (i.e. 7 mg/kg twice daily) to 42 mg/kg/day (i.e 21 mg/kg/day twice daily);
* Children ≥ 6 months to < 4 years:20 mg/kg/day (i.e. 10 mg/kg twice daily) to 60 mg/kg/day (i.e 30 mg/kg/day twice daily).

The first intravenous (IV) infusion was to be administered 12 hours after the last oral dose of levetiracetam.

For children not taking levetiracetam oral solution prior to entering the study, the intravenous (IV) dose will correspond to their age and weight as follows:

* Children ≥ 1 month to < 6 months: 14 mg/kg/day (i.e. 7 mg/kg twice daily).
* Children ≥ 6 months to < 4 years: 20 mg/kg/day (i.e. 10 mg/kg twice daily).

However, when necessary for the safety of the subject or when the investigator deemed it appropriate the levetiracetam intravenous (LEV IV) dose could be modified after one day.

Subjects were hospitalized for the duration of the levetiracetam intravenous (LEV IV) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 1 month and 4 years of age, inclusive
* The subject suffers from epilepsy (except status epilepticus)
* The subject is requiring levetiracetam IV treatment in place of oral therapy for a short period of time

Exclusion Criteria:

* The subject has difficult venous accessibility
* History of status epilepticus during the 3 months prior to Screening
* The subject is on felbamate with less than 18 months continuous exposure before Screening.
* The subject presents with current depressive symptoms, current suicidal ideation and/or behavior.

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (23):
- United States (6):
  - San Diego, California
  - Buffalo, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Richmond, Virginia
- Belgium (2):
  - Ghent
  - Leuven
- France (4):
  - Amiens
  - Lille
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (3):
  - Heidelberg
  - Kehl
  - Kiel
- Mexico (6):
  - Torreón, Coahuila
  - Puebla City, CP
  - Aguascalientes
  - Guadalajara
  - Mexico City
  - Puebla City
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir

REFERENCES:
- [Result] Weinstock A, Ruiz M, Gerard D, Toublanc N, Stockis A, Farooq O, Dilley D, Karmon Y, Elgie MJ, Schiemann-Delgado J. Prospective Open-Label, Single-Arm, Multicenter, Safety, Tolerability, and Pharmacokinetic Studies of Intravenous Levetiracetam in Children With Epilepsy. J Child Neurol. 2013 Nov;28(11):1423-1429. doi: 10.1177/0883073813480241. Epub 2013 Mar 26. PMID 23533164
- See also: FDA Safety Alerts and Links — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from sites in the United States, Belgium, Germany, France, Mexico, and Turkey. The study began in May 2008 and continued until March 2010, with the last subject's visit occurring in March of 2010.
Pre-assignment Details: Participant Flow refers to the Intent-to-treat (ITT) Population, consisting of all subjects who received at least 1 dose of study medication.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 19 (Of the 23 subjects screened, 19 were enrolled into the study and received levetiracetam IV (LEV IV).)
Completed | 16
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Other: Unable to obtain IV & PK samples | 1
Not completed — Other: IV dose needed to be changed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.59 (1.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 7
  Mexico | 8
  Belgium | 1
  Turkey | 2
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-Emergent Adverse Event (TEAE) During the Treatment Period (up to 4 Days)
Time Frame: Treatment period (up to 4 days)
Population: All 19 subjects enrolled in the study were included in the Intent to Treat (ITT) population and are included in this analysis.
Measure: Number; unit: Subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 19
Subjects | 12

2. Secondary Outcome: Number of Subjects Who Received High-dose Levetiracetam Intravenous (LEV IV) (More Than 28 mg/kg/Day for Subjects <6 Months; >40mg/kg/Day for Subjects ≥6 Months) During the Treatment Period (up to 4 Days)
Time Frame: Treatment period (up to 4 days)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 19
Subjects | 6

3. Secondary Outcome: Number of Consecutive Levetiracetam Intravenous (LEV IV) Doses Received
Time Frame: Treatment period (up to 4 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Consecutive doses
Arm/Group | Levetiracetam
Number analyzed (Participants) | 19
Consecutive doses | 2.89 (1.41)

ADVERSE EVENTS:
Time Frame: Up to 4 days
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=19)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (3)
ABDOMINAL SEPSIS (Infections and infestations) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 (2)
CONVULSION (Nervous system disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=19)
BRADYCARDIA (Cardiac disorders) | 1 (1)
EYE SWELLING (Eye disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
PYREXIA (General disorders) | 2 (2)
IRRITABILITY (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PUNCTURE SITE PAIN (General disorders) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1)
ELECTROENCEPHALOGRAM (Investigations) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (3)
DROOLING (Nervous system disorders) | 1 (1)
MYOCLONIC EPILEPSY (Nervous system disorders) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1)
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.